CLINICAL TRIAL: NCT05091372
Title: Minimal Residual Disease Guided Maintenance Therapy With Belantamab Mafodotin and Lenalidomide After Autologous Hematopoietic Cell Transplantation in Patients With Newly Diagnosed Multiple Myeloma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0201; NCI-2021-11334 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2021-10-12; First posted 2021-10-25 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Myeloma Multiple
MeSH Terms: conditions — Multiple Myeloma | interventions — belantamab mafodotin; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Belantamab mafodotin (Experimental): belantamab mafodotin by vein over about 30 minutes on Day 1 of each cycle
  Interventions: Drug: Belantamab mafodotin
- Lenalidomide (Experimental): lenalidomide by mouth every day of each cycle
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Belantamab mafodotin — Belantamab Mafodotin
  Belantamab mafodotin dose levels:
  Dose level -2 = 1.4 mg/kg IV every 12 weeks Dose level -1 = 1.9 mg/kg IV every 12 weeks Dose level 0 = 1.9 mg/kg IV every 8 weeks
  Cycles 1 - 6:
  All patients will start at dose level 0.
  Cycles 7 and onwards*:
  Patients previously on dose level 0 (1.9 mg/kg IV every 8 weeks) will change to dose level -1 (1.9 mg/kg IV every 12 weeks) Patients previously on dose level -1 (1.9 mg/kg IV every 12 weeks) will continue at the same dose level.
  Patients previously on dose level -2 (1.4 mg/kg IV every 12 weeks) will continue at the same dose level.
  *Reduction to a lower dose level is allowed in case of development of adverse effects or poor tolerance as determined by the treating physician.
  Arms: Belantamab mafodotin
Drug: Lenalidomide — Lenalidomide dose levels:
  Dose level 0 (starting dose): Lenalidomide 10 mg/day PO continuously. Dose level -1: Lenalidomide 10 mg/day PO. One week off after every three weeks of treatment.
  Dose level -2: Lenalidomide 5 mg/day PO. One week off after every three weeks of treatment.
  Other Names: CC-5013; Revlimid™
  Arms: Lenalidomide

SUMMARY:
To increase the conversion rate from MRD-positive to MRD-negative CR in patients with newly diagnosed multiple myeloma (NDMM) receiving post-transplant maintenance therapy with belantamab mafodotin plus lenalidomide.

DETAILED DESCRIPTION:
Primary Objective:

-To increase the conversion rate from MRD-positive to MRD-negative CR in patients with newly diagnosed multiple myeloma (NDMM) receiving post-transplant maintenance therapy with belantamab mafodotin plus lenalidomide.

Secondary Objectives:

* To determine the safety and tolerability of belantamab mafodotin plus lenalidomide maintenance therapy after auto-HCT.
* To increase the overall MRD-negative CR rate in patients with NDMM receiving post-auto-HCT maintenance therapy with belantamab mafodotin plus lenalidomide.
* To determine the PFS and OS in patients who discontinue maintenance therapy after achieving sustained MRD-negative CR. Sustained MRD-negative CR is defined as MRD-negative status in two assessments, at least 1-year apart, without any MRD-positive status in between.
* To determine the PFS with belantamab mafodotin plus lenalidomide maintenance therapy after auto-HCT in patients with NDMM.
* To determine the OS with belantamab mafodotin plus lenalidomide maintenance therapy after auto-HCT in patients with NDMMM.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed multiple myeloma status post 1st auto-HCT (day 60 - 180 post-transplant).
* Disease status (MRD positive or negative), partial response, or better.
* Age > 18-year and 75-year. Non-English speaking patients are eligible.
* Karnofsky performance status 70 (Appendix A.).
* Adequate organ function (Please see Table 2. below). Participant agrees to not donate blood while taking lenalidomide and for 28 days after stopping lenalidomide.
* Patient agrees to enroll in the lenalidomide REMS program.
* Woman of child-bearing potential (WOCPB) must abstain from hetersosexual sexual contact or agrees to use a contraceptive method that is highly effective (with a failure rate of <1% per year), preferably with low user dependency (as described in Appendix C), plus one additional effective method at least 28 days before starting therapy (for lenalidomide), during the intervention period, at least 28 days after the last dose of lenalidomide and at least 4 months after the last dose of belantamab mafodotin, and agrees not to donate eggs (ova, oocytes) for reproduction during this period. The investigator should evaluate the effectiveness of the contraceptive method in relation to the first dose of the study intervention.

A WOCBP must have a negative highly sensitive serum pregnancy test (as required by local regulations) within 10-14 days and also within 24 hours before the first dose of the study intervention.

Nonchildbearing potential is defined as follows (by other than medical reasons):

* ≥ 45 years of age and has not had menses for >1 year.
* Patients who have been amenorrhoeic for <2 years without a history of a hysterectomy and oophorectomy must have a follicle-stimulating hormone value in the postmenopausal range upon screening evaluation.
* Post-hysterectomy, post-bilateral oophorectomy, or post-tubal ligation. 9. Male participant agrees to contraceptive use that should be consistent with institutional guidelines regarding the methods of contraception for those participating in clinical studies.

Male participants are eligible to participate if they agree to the following during the intervention period and for 6 months after the last dose of study treatment to allow for clearance of any altered sperm:

• Refrain from donating sperm during treatment (including dose interruptions) and for 4 weeks after their last dose of lenalidomide.

PLUS, either:

• Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent.

OR Must agree to use contraception/barrier as detailed in Appendix C.

• All prior auto-HCT- related toxicities (defined by National Cancer Institute - Common Toxicity Criteria for Adverse Events (NCI-CTCAE), version 5 must be ≤ Grade 1 at the time of enrollment except for alopecia, fatigue, and amenorrhea.

Exclusion Criteria:

* History of progressive disease at any time before starting maintenance.
* Patients with smoldering MM (IMWG criteria, Appendix F.).
* Patients with plasma cell leukemia.
* Patients with non-secretory MM (no measurable disease on electrophoresis and immunofixation). Patients with a measurable disease on PET scan or bone marrow will be eligible.
* Participant must not have current unstable liver or biliary disease defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia due to underlying liver disease (serum albumin < 3gm/dL), esophageal or gastric varices, persistent jaundice, or cirrhosis. Note: Stable non-cirrhotic chronic liver disease (including Gilbert's syndrome or asymptomatic gallstones) or hepatobiliary involvement of malignancy is acceptable if otherwise meets entry criteria
* Participant must not have presence of active renal condition (infection, requirement for dialysis or any other condition that could affect participant's safety). Participants with isolated proteinuria resulting from MM are eligible, provided they fulfil inclusion criteria.
* Current corneal or epithelial disease (except mild punctate keratopathy; see Appendix E.).
* Participant must not use contact lenses while participating in this study.
* Participant must not have used an investigational drug or approved systemic anti-myeloma therapy (including systemic steroids) within 14 days or five half-lives, whichever is shorter, preceding the first dose of study drug.
* Participant must not have received prior treatment with a monoclonal antibody within 30 days of receiving the first dose of study drugs.
* Participant must not have had major surgery ≤ 4 weeks before initiating study treatment.
* The participant must not have any evidence of active mucosal or internal bleeding.
* Participant must not have known immediate or delayed hypersensitivity reaction or idiosyncratic reactions to belantamab mafodotin or drugs chemically related to belantamab mafodotin, or any of the components of the study treatment.
* Participant must not have an active infection requiring treatment.
* Participant must not have evidence of cardiovascular risk, including any of the following:

  1. Evidence of current clinically significant uncontrolled arrhythmias, including clinically significant ECG abnormalities such as 2nd degree (Mobitz Type II) or 3rd degree atrioventricular (AV) block.
  2. History of myocardial infarction, acute coronary syndromes (including unstable angina), coronary angioplasty, or stenting or bypass grafting within three (3) months of screening.
  3. Class III or IV heart failure as defined by the New York Heart Association functional classification system.16
  4. Uncontrolled hypertension (blood pressure that remains above goal despite the concurrent use of three antihypertensive drug classes).
* Participant must not have known HIV infection.
* Patients will Hepatitis B will be excluded unless the following criteria can be met (Please, also see Appendix B):

Serology Screening HbcAb+, HbsAg- • HBV DNA undetectable HBsAg+ at screen or within 3 months prior to first dose • HBV DNA undetectable

* Highly effective antiviral treatment started at least 4 weeks prior to first dose of study treatment
* Baseline imaging per protocol
* Participants with cirrhosis are excluded

Note: presence of Hep B surface antibody (HBsAb) indicating previous vaccination will not exclude a participant.

* Positive hepatitis C antibody test result or positive hepatitis C RNA test result at screening or within 3 months prior to first dose of study treatment unless the participant can meet the following criteria (Please, also see Appendix B):

  * RNA test negative
  * Successful anti-viral treatment (usually 8 weeks duration) is required, followed by a negative HCV RNA test after a washout period of at least 4 weeks.
* Participant must not have invasive malignancies other than disease under study, unless the second malignancy has been medically stable for at least 2 years and, in the opinion of the principal investigators, will not affect the evaluation of the effects of clinical trial treatments on the currently targeted malignancy. Participants with curatively treated non-melanoma skin cancer may be enrolled without a 2-year restriction.
* Participants must not be pregnant or lactating.
* Patients with cognitive impairments and/or any serious unstable pre-existing medical condition or psychiatric disorder that can interfere with safety or with obtaining informed consent or compliance with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Conversion rate from MRD-positive to MRD-negative CR in patients with newly diagnosed multiple myeloma (NDMM) receiving post-transplant maintenance therapy with belantamab mafodotin plus lenalidomide. | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Qaiser Bashir, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Mohan M, Gundarlapalli S, Szabo A, Yarlagadda N, Kakadia S, Konda M, Jillella A, Fnu A, Ogunsesan Y, Yarlagadda L, Thalambedu N, Munawar H, Graziutti M, Al Hadidi S, Alapat D, Thanendrarajan S, Zangari M, van Rhee F, Schinke C. Tandem autologous stem cell transplantation in patients with persistent bone marrow minimal residual disease after first transplantation in multiple myeloma. Am J Hematol. 2022 Jun 1;97(6):E195-E198. doi: 10.1002/ajh.26530. Epub 2022 Mar 21. No abstract available. PMID 35285981
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2025-03-04): https://cdn.clinicaltrials.gov/large-docs/72/NCT05091372/ICF_001.pdf